CLINICAL TRIAL: NCT07156448
Title: Effectiveness of Exercise Intervention on Physical Function, Psychological Health, Quality of Life, and Spiritual Well-Being in Hospitalized Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE21145B; TCVGH-1107402B (Other: Taichung Veterans General Hospital, Taiwan)
Record Dates: First submitted 2025-08-20; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hospitalization; Aged 65 Years or Older; Activities of Daily Living; Depression; Quality of Life; Spirituality
Keywords: Exercise intervention; Physical function; Mobility; Timed Up and Go; Barthel Index; Functional Reach Test; Handgrip strength; Geriatric Depression Scale; EQ-5D-3L; EQ-VAS; Spiritual Index of Well-Being; Spiritual well-being; Internal medicine ward; Older patients
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received the exercise program, or the control group, which received usual care. Both groups were assessed at baseline and after the intervention
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts were blinded to group allocation to minimize assessment and analysis bias. Participants and care providers were not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (Experimental): Participants received a structured exercise program during hospitalization, including resistance training, stretching, and walking, delivered five times per week for 30 minutes per session.
  Interventions: Behavioral: Multicomponent Exercise Program
- Control Group (No Intervention): Participants received usual hospital care without additional structured exercise intervention.

INTERVENTIONS:
Behavioral: Multicomponent Exercise Program — Participants in the intervention group received a structured, multicomponent exercise program consisting of resistance training, stretching, and walking. The program began on the second day of hospitalization and continued until discharge, with a frequency of five sessions per week. Each session lasted approximately 30 minutes, including about 20 minutes of resistance and stretching exercises targeting major muscle groups through functional movements (e.g., sit-to-stand, leg flexion-extension) and flexibility exercises for the upper arms, back, and posterior legs, performed in 2 to 3 sets of 8 to 12 repetitions. Each session also incorporated approximately 10 minutes of walking, with intensity adjusted according to individual tolerance.
  Arms: Exercise Intervention Group

SUMMARY:
This study aimed to evaluate the effects of a structured exercise program on physical function, psychological well-being, quality of life, and spiritual well-being in hospitalized older adults. A total of 100 inpatients aged 65 years or older were assigned to either an intervention group or a control group. The intervention group participated in a multicomponent exercise program during hospitalization, including resistance training, stretching, and walking, while the control group received routine care. Assessments were performed before and after the intervention using physical performance tests, questionnaires, and well-being scales. The goal is to determine whether such a program can improve mobility, daily living independence, mood, and overall well-being in older patients during hospitalization.

DETAILED DESCRIPTION:
This single-center, parallel-group randomized controlled trial investigated the effects of a structured exercise program on multiple dimensions of health in hospitalized older adults. Eligible participants were adults aged ≥65 years, admitted from the emergency department to two internal medicine wards in a teaching hospital in central Taiwan, able to communicate, capable of standing and walking (with or without assistive devices), and willing to participate in the program.

Participants in the intervention group received a structured, multicomponent exercise program consisting of resistance training, stretching, and walking. The program began on the second day of hospitalization and continued until discharge, with a frequency of five sessions per week. Each session lasted approximately 30 minutes, including about 20 minutes of resistance and stretching exercises targeting major muscle groups through functional movements (e.g., sit-to-stand, leg flexion-extension) and flexibility exercises for the upper arms, back, and posterior legs, performed in 2 to 3 sets of 8 to 12 repetitions. Each session also incorporated approximately 10 minutes of walking, with intensity adjusted according to individual tolerance. All sessions were supervised by trained nurses or physical therapists to ensure correct performance and safety.

The control group received routine inpatient care without structured exercise.

Primary outcomes included measures of physical function (Timed Up and Go test, 6-meter walk test, Functional Reach Test, Handgrip strength, and Barthel Index) and psychological health (5-item Geriatric Depression Scale). Secondary outcomes included quality of life (EQ-5D-3L, EQ Visual Analogue Scale) and spiritual well-being (Spiritual Index of Well-Being). All assessments were conducted at baseline (admission) and before discharge by trained assessors blinded to group allocation.

The study aimed to determine whether implementing a structured exercise program during hospitalization could improve multidimensional health outcomes, and to provide evidence for integrating holistic, non-pharmacological interventions into geriatric inpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Able to communicate
* Capable of standing and walking (with or without assistive devices)
* Willing to participate in both the study and the exercise intervention

Exclusion Criteria:

* Impaired consciousness
* Acute inflammatory conditions (e.g., gout, acute myocardial infarction, unstable angina, heart failure)
* Physician-ordered activity restrictions at admission
* Diagnosed psychiatric disorders or history of epilepsy
* Severe disability requiring total assistance in daily life

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Assesses mobility and balance by timing the participant as they rise from a chair, walk 3 meters, turn, walk back, and sit down. Time recorded in seconds; shorter times indicate better performance.
6-meter walk test (6MWT) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  6-meter walk test (6MWT), which measured gait speed, with speeds <1.0 m/s suggesting reduced independence
Functional Reach Test (FRT) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Assesses dynamic balance by measuring the maximum forward reach distance beyond arm's length while standing, in centimeters. A reach <15 cm indicates higher fall risk.
Handgrip strength (HGS) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Measures maximal grip force using a handheld dynamometer, recorded in kilograms. Cut-offs: <26 kg (men) and <18 kg (women) indicate sarcopenia.
Barthel Index (BI) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Assesses independence in activities of daily living (ADL) on a scale of 0-100; higher scores indicate better function.
5-item Geriatric Depression Scale (GDS-5) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Self-report questionnaire assessing depressive symptoms. Scores ≥2 suggest probable depression.

SECONDARY OUTCOMES:
EuroQol 5-Dimension 3-Level (EQ-5D-3L) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Assesses five health domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) on three severity levels.
EuroQol Visual Analogue Scale (EQ-VAS) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  Self-rated health status from 0 (worst imaginable) to 100 (best imaginable).
Spiritual Index of Well-Being (SIWB) | Baseline (Day 2 of hospitalization) and at discharge (within 24 hours prior to hospital discharge, average length of stay 10 days)
  12-item questionnaire with two subscales (self-efficacy and life scheme), scored on a 5-point Likert scale. Higher scores reflect poorer spiritual well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results, including baseline characteristics and all primary and secondary outcome measures, will be shared. A data dictionary will be provided to describe variable definitions. Data will be available upon reasonable request after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication and ending 5 years thereafter
Access Criteria: Researchers must submit a methodologically sound research proposal and sign a Data Use Agreement. Requests will be reviewed by the principal investigator to ensure compliance with ethical and legal requirements.